CLINICAL TRIAL: NCT02699658
Title: Population Pharmacokinetics and Pharmacodynamics Modeling to Optimize Dosage Regimen of Levofloxacin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sutep Jaruratanasirikul, Prince of Songkla University, Prince of Songkla University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Levo-57-356141
Record Dates: First submitted 2016-02-24; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Healthy Volunteers
Keywords: levofloxacin; population pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- levofloxacin in healthy (Experimental)
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
Levofloxacin, a fluoroquinolone antibiotic, is the optical S-(-) isomer of ofloxacin with a broad spectrum of activity. In common with other fluoroquinolones, the main pharmacokinetic/pharmacodynamic (PK/PD) index that correlates with its therapeutic efficacy is the area under the plasma time-concentration curve/the minimum inhibitory concentration ratios.

The aims of the study were to:

1. reveal the population pharmacokinetics, and
2. assess the efficacy of various dosage regimens in achieving the probability of target attainment (PTA) and the cumulative fraction of response (CFR) of levofloxacin when oral levofloxacin was prescribed as the switching therapy after intravenous levofloxacin treatment.

The study was conducted in 45 healthy volunteers. Each subject received one 500 mg tablet of levofloxacin, after which PK studies were carried out, using a Monte Carlo simulation to determine the PTA. By referral to the EUCAST MIC distributions database, the dosage regimens were predicted to achieve CFR greater than or equal to 90%.

ELIGIBILITY:
Inclusion:

* normal hematologic
* normal hepatic
* normal renal functions
* non-smoking
* non-alcoholic
* non-obese

Exclusion:

* pregnant or lactating women
* any chronic medications

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
concentration of levofloxacin in plasma | up to 2 week after blood collection

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand